CLINICAL TRIAL: NCT01141985
Title: Evaluation Of A New Disposable Contact Lens Patient Interface For The Lensx Laser In Cataract And Corneal Surgery
Brief Title: New Disposable Contact Lens Patient Interface For The Lensx Laser
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: LenSx Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CPT-001h
Record Dates: First submitted 2010-06-04; First posted 2010-06-11 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Cataract; Corneal Disease
Keywords: cataract; cornea; keratoplasty
MeSH Terms: conditions — Cataract; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated (Other): This is a single arm study.
  Interventions: Device: LenSx Laser modified disposable contact lens

INTERVENTIONS:
Device: LenSx Laser modified disposable contact lens — Modified Disposable Contact Lens Patient Interface: Like the current disposable contact lens, a single unit is used for each procedure only once, and is then discarded. It is similarly mounted onto the distal end of the system's focusing objective and serves as a sterile barrier between the patient and the laser. In place of a separate suction ring that is used in the current contact lens, the modified contact lens has an integrated suction ring and curved applanation surface. These features result in significantly lower elevation of intraocular pressure and significantly easier application by the surgeon in preliminary testing. Identical to the current contact lens, the suction ring is applied around the patient's limbus and mild suction is applied to stabilize the eye.

SUMMARY:
The objective of this study is to evaluate the ease of use of a modified, disposable contact lens and suction ring assembly.

DETAILED DESCRIPTION:
This will be a prospective, single center clinical trial of up to 300 consecutive eyes of subjects scheduled to undergo ocular surgery requiring an initial incision, specifically, cataract surgery. Subjects will be screened for eligibility. Eligible subjects will be examined preoperatively to establish a baseline for ocular condition.

Subjects will undergo unilateral cataract surgery using the LenSx Laser for one or a combination of the following laser procedures: anterior capsulotomy, laser lens phacofragmentation and corneal incision with implantation of an intraocular lens (IOL). Surgeon and staff comments will be solicited for ergonomic and packaging features of the new disposable contact lens. Subjects will be evaluated intraoperatively to assess comfort of the new disposable contact lens, as well as the completion of anterior capsulotomy, laser lens phacofragmentation and completion of corneal incisions. All patients will be evaluated postoperatively at one day, one week and 1 month to follow the condition of the surgical eye. Further follow up can be performed at the discretion of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens implantation in at least 1 eye.
2. Subjects must be at least 24 years of age.
3. Subjects must be willing and able to return for scheduled follow-up examinations.
4. Subjects must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

1. Subjects with corneal disease or pathology that precludes applanation of the cornea or transmission of laser wavelength or distortion of laser light are excluded.
2. Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally are excluded.
3. Subjects with residual, recurrent, active ocular or eyelid disease, including any corneal abnormality (for example, recurrent corneal erosion, severe basement membrane disease) in either eye are excluded.
4. Subjects with a history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP>21 mm Hg in either eye are excluded.
5. Subjects with known lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
6. Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye are excluded.
7. Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study are excluded.
8. Subjects with known sensitivity to planned study concomitant medications are excluded.
9. Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation are excluded
10. Subjects presenting any contraindications to cataract surgery are excluded.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Disposable contact lens successfully applied to the eye | Intraoperative (Day 0)
  Was the Contact Lens successfully applied to the eye? Yes or No.

SECONDARY OUTCOMES:
Surgical evaluation of Corneal Incision | Intraoperative (Day 0)
  Was the corneal incision complete?
Standard Outcomes Measurements | Pre-operative (Day -60 to Day -1)
  Standard measurements of Visual Acuity, Manifest Refraction, Slit Lamp Examination, Fundus Examination, Intraocular pressure, Complications and Adverse Events
Surgical evaluation of capsulotomy | Intraoperative (Day 0)
  Was capsulotomy complete? Yes or No.
Surgical evaluation of fragmentation | Intraoperative (Day 0)
  Was lens fragmentation complete? Yes or No.
Standard outcomes measurement | 1 week (5 to 10 days post operative)
  Standard measurements of Visual Acuity, Manifest Refraction, Slit Lamp Examination, Fundus Examination, Intraocular pressure, Complications and Adverse Events
Standard outcomes measurement | 1 day (24 to 48 hours postoperative)
  Standard measurements of Visual Acuity, Manifest Refraction, Slit Lamp Examination, Fundus Examination, Intraocular pressure, Complications and Adverse Events
Standard outcomes measurement | 1 month (21 to 42 days postoperative)
  Standard measurements of Visual Acuity, Manifest Refraction, Slit Lamp Examination, Fundus Examination, Intraocular pressure, Complications and Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Slade, MD, Principal Investigator — Slade and Baker Vision Center
Locations (1):
- Slade and Baker Vision Center, Houston, Texas, United States